CLINICAL TRIAL: NCT00571220
Title: Mechanisms of Diabetes Control After Weight Loss Surgery
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK67561 (completed); R01DK067561 (NIH)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Gastric Bypass Surgery; Obesity
Keywords: gastric bypass; diabetes; obesity; diet-induced weight loss; incretin levels (GLP-1,GIP); incretin effect
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gastric bypass surgery: Surgical group of obese patients with type 2 diabetes undergoing gastric bypass surgery
  Interventions: Procedure: gastric bypass surgery
- Diet induced weight loss: Diet group of obese patient with type 2 diabetes, matched with the surgical group for diabetes duration, diabetes control (HbA1C), BMI, age.
  Interventions: Other: Diet induced weight loss

INTERVENTIONS:
Procedure: gastric bypass surgery — weight loss bariatric surgery
  Groups: Gastric bypass surgery
Other: Diet induced weight loss — low calorie diet with meal replacements. weekly outpatient visits with nutritionist.
  Groups: Diet induced weight loss

SUMMARY:
Obesity and type 2 diabetes (T2DM) are increasing in the US. One third of patients seeking bariatric surgery have T2DM. Although all surgeries result in significant weight loss and often 'cure' the T2DM, the rapid onset and the magnitude of the benefits of gastric bypass (GBP) on T2DM has thus far baffled clinical scientists. Limited data suggest that the improvement in T2DM after GBP occurs very rapidly, and may not be wholly accounted for by weight loss. Secretion of incretins (gut peptides secreted in response to meals which enhance insulin secretion) is impaired in T2DM and improves after GBP, possibly due to the specific anatomical changes after this surgery. While some determinants of impaired insulin secretion, such as glucotoxicity, improve equally after diet or surgical weight loss, the improvement in the incretin effect after GBP might be specific to this surgery. The aim of this study is to determine whether the magnitude of the incretin effect on insulin secretion is greater after GBP than after an equivalent diet-induced weight loss. We will compare, in obese patients with diabetes, randomized to very low calorie diet or to GBP, the effect of an equivalent weight loss on the incretin effect (difference in insulin secretion after comparable oral and intravenous (IV) glucose loads). As more obese diabetic patients undergo GBP, understanding the mechanisms that produce improvement in their diabetes is increasingly important.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese with type 2 diabetes candidates and being evaluated at our institution for bariatric surgery (group1); morbidly obese patients with type 2 diabetes who want to lose weight by diet.

Exclusion Criteria:

* any condition that would be contra-indicated for bariatric surgery (ex:unstable angina)
* diabetes treated by insulin, thiazolidinediones (TZD), exenatide, DPP-IV inhibitors
* HbA1C > 8%

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Morbidly obese patients with type 2 diabetes of less than 5 years duration
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in incretin | One month
  Change in incretin (gastric inhibitory peptide [GIP] and glucagon-like peptide-1 [GLP-1])

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St Luke's Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Result] Laferrere B, Heshka S, Wang K, Khan Y, McGinty J, Teixeira J, Hart AB, Olivan B. Incretin levels and effect are markedly enhanced 1 month after Roux-en-Y gastric bypass surgery in obese patients with type 2 diabetes. Diabetes Care. 2007 Jul;30(7):1709-16. doi: 10.2337/dc06-1549. Epub 2007 Apr 6. PMID 17416796
- [Derived] Dutia R, Brakoniecki K, Bunker P, Paultre F, Homel P, Carpentier AC, McGinty J, Laferrere B. Limited recovery of beta-cell function after gastric bypass despite clinical diabetes remission. Diabetes. 2014 Apr;63(4):1214-23. doi: 10.2337/db13-1176. Epub 2013 Dec 2. PMID 24296713
- [Derived] Laferrere B, Swerdlow N, Bawa B, Arias S, Bose M, Olivan B, Teixeira J, McGinty J, Rother KI. Rise of oxyntomodulin in response to oral glucose after gastric bypass surgery in patients with type 2 diabetes. J Clin Endocrinol Metab. 2010 Aug;95(8):4072-6. doi: 10.1210/jc.2009-2767. Epub 2010 May 25. PMID 20501690